CLINICAL TRIAL: NCT03281941
Title: ToAST: Investigating the Effect of Bronchial Thermoplasty on Cough in Patients With Severe Asthma
Brief Title: ToAST:Investigating the Effect of Bronchial Thermoplasty on Cough in Patients With Severe Asthma
Acronym: ToAST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Health Service, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Ran Wang, Dr Ran Wang (Chief Investigator); Professor Jacky Smith (PI), National Health Service, United Kingdom
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NHSUK
Record Dates: First submitted 2017-08-22; First posted 2017-09-13 (Actual); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Asthma Chronic, Cough
MeSH Terms: conditions — Cough

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients without BT (Other)
  Interventions: Other: Inhaled capsaicin cough challenge
- Post BT (Other)
  Interventions: Other: Inhaled capsaicin cough challenge

INTERVENTIONS:
Other: Inhaled capsaicin cough challenge

SUMMARY:
ToAST study is a pilot study aiming to establish the safety profile of using inhaled capsaicin challenge in patients with severe asthma. The investigators will also explore the differences in cough symptoms and threshold in patients with and without bronchial thermoplasty.

DETAILED DESCRIPTION:
ToAST is designed as a two-visit observational study. During visit 1, written consent and measurements of baseline asthma characteristics were completed; history and examination, questionnaires (Asthma Control Questionnaires and Leicester Cough Questionnaire, and basic lung physiological assessment were performed.

At the end of visit 1, a cough monitor was attached to the subject to monitor cough frequency for the next 24 hours and this was returned at visit 2.

Visit 2 followed within two weeks after visit 1, during which a full dose capsaicin cough challenge was performed. Emergency contact details were given towards end of visit 2 should any adverse events occur.

Telephone call within 48 hours, Day 3 and Day 7: The purpose of these phone calls was to ensure that the patient had not developed any adverse effects to the capsaicin challenge.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18
* Person with an established diagnosis of severe asthma
* All patients should be on British Thoracic Society (BTS) steps 4 or 5
* Patients who have had bronchial thermoplasty (BT) should be at least 2 months after their treatment
* Historical evidence of one of the following:
* Airway reversibility to a short acting beta-2 agonist of ≥12%
* Bronchial hyper-responsiveness (PC20<8mg/ml)
* Fractional exhaled nitric oxide ≥50ppb
* Peak flow variability >8%
* Raised serum (≥0.45) or sputum eosinophilia (>3%)
* Variability in spirometry over 24 months of >20%

Exclusion Criteria:

* Unable to give informed consent
* FEV1<50% predicted or < 1 litre
* Known allergy or intolerance to capsaicin
* Symptoms of upper respiratory tract infection in the last 1 month which have not resolved.
* Lower respiratory tract infection or pneumonia in the last 6 weeks.
* Current smoker or ex-smoker with ≥10 pack year smoking history, abstinence of ≤6 months
* Asthma exacerbation in the previous month requiring an increase or starting of an ICS or OCS
* Subject has changed asthma medication within the past 4 weeks prior to screening
* A previous asthma exacerbation requiring Intensive Care Unit (ICU) admission.
* Significant other pulmonary disorders as the major diagnosis, in particular: pulmonary embolism, pulmonary hypertension, interstitial lung disease, lung cancer, cystic fibrosis, emphysema or bronchiectasis.
* Evidence of vocal cord dysfunction
* Pregnancy or breast-feeding
* Use of ACE inhibitors
* Any centrally acting medication which in the view of the investigator could alter the sensitivity of the cough reflex*
* History of psychiatric illness, drug or alcohol abuse which may interfere in the participation of the trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-08-06 (Actual); Primary Completion 2018-02-01 (Estimated); Study Completion 2018-02-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants who has had significant fall in FEV1 (defined as >20%) within the challenge period | Through study completion, an average of 6 months
  By measuring spirometry immediately before and after challenge
Number of participants who require bronchodilator treatment during capsaicin challenge period | Through study completion, an average of 6 months
  Defined as rescue medications - 2 puffs of salbutamol inhaler via spacer

SECONDARY OUTCOMES:
Change in %FEV1 predicted during capsaicin challenge period in all subjects | Through study completion, an average of 6 months
  By measuring spirometry immediately before and after challenge
The tolerability of inhaled capsaicin in severe asthma | Through study completion, an average of 6 months
  By exploring the pattern of termination of challenge in severe asthma
The number of adverse events in all subjects during and after capsaicin evoked cough challenge | Through study completion, an average of 6 months
  by follow up phone calls at 48 hours, 3 days and 7 days to assess AE and SAE
Degree of breathlessness during capsaicin challenge period assessed by using modified Borg scale (mBorg). | Through study completion, an average of 6 months
  By calculating Borg immediately before and after challenge to assess level of breathlessness.
Degree of breathlessness during capsaicin challenge period assessed by using dysnoea Visual Analogue Score (dVAS). | Through study completion, an average of 6 months
  By calculating dVAS immediately before and after challenge to assess level of breathlessness.
Differences in capsaicin dose response curves (Maximum cough response evoked by any concentration of capsaicin- Emax and Capsaicin dose inducing half-maximal response - ED50) between subjects who have had BT versus those have not | Through study completion, an average of 6 months
  by comparing post-BT and no-BT patients
The differences in 24-hour cough frequency between patients who have had BT and those who have not. | Through study completion, an average of 6 months
  by comparing post-BT and no-BT patients
The differences in Leicester cough questionnaire (LCQ) between patients who have had BT and those who have not. | Through study completion, an average of 6 months
  by comparing post-BT and no-BT patients
The differences in asthma control questionnaire(ACQ) between patients who have had BT and those who have not. | Through study completion, an average of 6 months
  by comparing post-BT and no-BT patients
The differences of the dose response curves in patients with severe asthma with existing data of capsaicin challenge in patients with healthy and mild/moderate asthma (in Emax and ED50). | Through study completion, an average of 6 months
  By comparing with existing data.

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of South Manchester, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided